CLINICAL TRIAL: NCT00109070
Title: A Phase III, Multicenter, Randomized, Active-Controlled Clinical Trial to Evaluate the Efficacy and Safety of rhuMAb VEGF (Bevacizumab) in Combination With Standard Chemotherapy in Subjects With Metastatic Colorectal Cancer
Brief Title: A Study to Evaluate Avastin in Combination With Standard Chemotherapy to Treat Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: AVF2107g; NCT00012233 (obsolete NCT alias)
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab

INTERVENTIONS:
Drug: Avastin (bevacizumab)

SUMMARY:
This is a multicenter, Phase III, randomized, active-controlled trial to evaluate the efficacy and safety of rhuMAb VEGF (Avastin) added to the standard first-line chemotherapy used to treat metastatic colorectal cancer. This trial will enroll approximately 900 subjects with histologically confirmed, previously untreated, bi-dimensionally measurable metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >=18 years
* Histologically confirmed colorectal carcinoma with evidence of metastases (i.e., by radiographic imaging or biopsy)
* Ability to tolerate CT contrast dye
* Bi-dimensionally measurable disease (minimum of two lesions)
* ECOG performance status of 0 or 1
* Use of an effective means of contraception in women of childbearing potential
* Life expectancy of >3 months
* Willingness and capability to be accessible for follow-up until death or study termination by Genentech

Exclusion Criteria:

* Prior chemotherapy other than adjuvant fluoropyrimidines in combination with leucovorin and/or levamisole
* Administration of adjuvant fluoropyrimidines in combination with leucovorin and/or levamisole completed <=12 months prior to Day 0
* Administration of fluoropyrimidines as a radiosensitizer during pelvic radiotherapy for rectal cancer completed <=12 months prior to Day 0
* Prior radiotherapy to a measurable, metastatic lesion(s) to be used to measure response
* Radiation therapy within 14 days prior to Day 0
* Prior biotherapy for colorectal cancer
* Evidence of clinically detectable ascites on Day 0
* Other invasive malignancies within 5 years prior to Day 0 (other than basal cell carcinoma of the skin)
* History or evidence upon physical examination of CNS disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke)
* Active infection requiring parenteral antibiotics on Day 0
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations within 7 days prior to Day 0
* Current or recent (within the 10 days prior to Day 0) use of full-dose oral or parenteral anticoagulants (except as required to maintain patency of preexisting, permanent indwelling IV catheters) or thrombolytic agent (for subjects receiving warfarin, international normalized ratio [INR] of <1.5; appropriate use of heparin should be discussed with the Medical Monitor)
* Chronic, daily treatment with aspirin (>325 mg/day) or nonsteroidal anti-inflammatory medications (of the kind known to inhibit platelet function at doses used to treat chronic inflammatory diseases)
* Pregnancy (positive pregnancy test) or lactation
* Proteinuria at baseline or clinically significant impairment of renal function
* Serious, nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Current or recent (within the 28 days prior to Day 0) participation in another experimental drug study
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year prior to Day 0
* Screening clinical laboratory values: *ANC of <1500/uL; *Platelet count of <75,000/uL; *INR of >=1.5; *Total bilirubin of >1.6 mg/dL; *AST or ALT >=5 times upper limit of normal for subjects with documented liver metastases (>2.5 times the upper limit of normal for subjects without evidence of liver metastases); *Serum creatinine of >2.0 mg/dL; *Hemoglobin of <9 gm/dL (may be transfused to maintain or exceed this level)
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2003-04 (Actual)

REFERENCES:
- [Result] Scappaticci FA, Skillings JR, Holden SN, Gerber HP, Miller K, Kabbinavar F, Bergsland E, Ngai J, Holmgren E, Wang J, Hurwitz H. Arterial thromboembolic events in patients with metastatic carcinoma treated with chemotherapy and bevacizumab. J Natl Cancer Inst. 2007 Aug 15;99(16):1232-9. doi: 10.1093/jnci/djm086. Epub 2007 Aug 8. PMID 17686822
- [Result] Kabbinavar FF, Wallace JF, Holmgren E, Yi J, Cella D, Yost KJ, Hurwitz HI. Health-related quality of life impact of bevacizumab when combined with irinotecan, 5-fluorouracil, and leucovorin or 5-fluorouracil and leucovorin for metastatic colorectal cancer. Oncologist. 2008 Sep;13(9):1021-9. doi: 10.1634/theoncologist.2008-0003. Epub 2008 Sep 5. PMID 18776057
- [Result] Grothey A, Hedrick EE, Mass RD, Sarkar S, Suzuki S, Ramanathan RK, Hurwitz HI, Goldberg RM, Sargent DJ. Response-independent survival benefit in metastatic colorectal cancer: a comparative analysis of N9741 and AVF2107. J Clin Oncol. 2008 Jan 10;26(2):183-9. doi: 10.1200/JCO.2007.13.8099. PMID 18182660
- [Result] Kabbinavar FF, Hurwitz HI, Yi J, Sarkar S, Rosen O. Addition of bevacizumab to fluorouracil-based first-line treatment of metastatic colorectal cancer: pooled analysis of cohorts of older patients from two randomized clinical trials. J Clin Oncol. 2009 Jan 10;27(2):199-205. doi: 10.1200/JCO.2008.17.7931. Epub 2008 Dec 8. PMID 19064978
- [Result] Lu JF, Bruno R, Eppler S, Novotny W, Lum B, Gaudreault J. Clinical pharmacokinetics of bevacizumab in patients with solid tumors. Cancer Chemother Pharmacol. 2008 Oct;62(5):779-86. doi: 10.1007/s00280-007-0664-8. Epub 2008 Jan 19. PMID 18205003
- [Result] Hurwitz HI, Yi J, Ince W, Novotny WF, Rosen O. The clinical benefit of bevacizumab in metastatic colorectal cancer is independent of K-ras mutation status: analysis of a phase III study of bevacizumab with chemotherapy in previously untreated metastatic colorectal cancer. Oncologist. 2009 Jan;14(1):22-8. doi: 10.1634/theoncologist.2008-0213. Epub 2009 Jan 14. PMID 19144677